CLINICAL TRIAL: NCT02313987
Title: The Impact of Endothelial Function-guided Therapy Compared to Usual Care on Major Adverse Cardiovascular Events in Patients With Chest Pain and Non-obstructive Coronary Artery Disease
Brief Title: Endothelial Function-guided Therapy Compared to Usual Care in Patients With NOCAD
Acronym: EndoGET
Status: Withdrawn | Type: Observational
Why Stopped: Study never began
Sponsor: Itamar-Medical, Israel (Industry)
Responsible Party: Sponsor
Other Study IDs: Endo-EndoGET-001
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Coronary Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- A-Usual care- Standard care for NOCAD: Subjects with non obstructive CAD (20-70% luminal diameter stenosis) and normal Endothelial function as defined by EndoScore.
  These subjects will receive the standard care usually provided in each facility for patients with NOCAD
- B1-Usual Care-Standard care for NOCAD: Subjects with non obstructive CAD (20-70% luminal diameter stenosis ) and abnormal Endothelial function as defined by EndoScore.
  These subjects will receive the standard care usually provided in each facility for patients with NOCAD. (Same care as Group A)
- B2- Endothelial function guid care: Subjects with non obstructive CAD and abnormal Endothelial function as defined by EndoScore.
  These subjects will receive the an Endothelial Function-guided Therapy.

SUMMARY:
The current study is designed to test the hypothesis that compared to conventional treatment; endothelial function-guided treatment reduces adverse cardiovascular events in patients with non-obstructive coronary artery disease documented at clinically indicated coronary angiography.

DETAILED DESCRIPTION:
Subjects with chest pain and non-obstructive coronary artery disease (20-70% luminal diameter narrowing) documented by coronary angiograms will be enrolled in the study 2 - 30 days following the coronary angiograms. Only subjects who have signed an Informed Consent Form and meet all of the eligibility criteria will be qualified for enrollment.

Following the baseline EndoPAT testing subjects will be divided into two groups by their EndoPAT (EndoScore) results:

1. Group A - normal EndoScore: Logarithmic value of RHI (Ln_RHI) >0.7
2. Group B - abnormal EndoScore: Ln_RHI ≤ 0.7 The subjects of Group B will be randomized in 1:1 ratio (by envelopes with randomization numbers at each site) to Group B1 who will be treated conventionally i.e., "usual care" by the site study team; and Group B2 who will be treated with "enhanced care".

Staff prescribing treatment regime for subjects in group A and B1 ("usual care") along with the subjects in these groups, will be blinded to the EndoScore value.

Subjects of all groups will return for 4 follow-up visits: 180±14days, 360±14days, 720±14days and 1080±14days (study end).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with chest pain and non-obstructive coronary artery disease documented by coronary angiography with 20-70% luminal diameter stenosis that does not justify coronary revascularization
* Stable subjects without evidence of prior MI/CABG/PTCA.
* Age 20 to 79 years
* Ability to understand the study procedures and provide written informed consent
* Willingness and ability to comply with the study and its scheduled visits and study procedures

Exclusion Criteria:

* Age below 20 over 79 years
* Subjects with documented MI, PTCA or CABG
* Unstable angina
* Any lesion > 20% luminal narrowing in the left main coronary artery
* Congestive heart failure, NYHA class II - IV
* Severe renal dysfunction, defined as an estimated glomerular filtration rate (eGFR calculated by MDRD) < 20 mL/min/1.73m2 at screening
* Uncontrolled hyperthyroidism or hypothyroidism as defined by thyroid stimulating hormone (TSH) , 1.0 time the lower limit of normal (LLN) or > 1.5 times the upper limit of normal (ULN), respectively, at screening
* Symptomatic peripheral artery disease
* History of drug or alcohol abuse
* Active liver disease or hepatic dysfunction, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) 2 times the ULN as determined by local laboratory analysis at screening
* Prior CVA or TIA
* Malignancy (except non-melanoma skin cancers, cervical in-situ carcinoma, breast ductal carcinoma in situ or stage 1 prostate carcinoma) with life expectancy of < 3 years
* Any planned surgery within 3 months after randomization
* Recipient of any major organ transplant (e.g., heart, lung, liver, bone marrow)
* Severe, concomitant non-cardiovascular disease that is expected to reduce life expectancy to less than 3 years
* Known, concerning active infection or major hematologic, renal, metabolic, gastrointestinal or endocrine dysfunction in the judgment of the investigator
* Currently enrolled in another investigational device or drug study, or less than 30 days since ending another investigational device or drug study(s), or receiving other investigational agent(s). Special clearance can be obtained from the Steering Committee for subjects enrolled in studies not conflicting with this protocol
* History or evidence of any other clinically significant disorder, condition or disease other than those outlined above that, in the opinion of the investigator may compromise the ability of the subject to give written informed consent, would pose a risk to the subject safety, or interfere with the study evaluation, procedures or completion
* Deformities of the digits of the upper extremities, which preclude adequate signal acquisition
* Subjects under the effect of short-acting NTG (3 hours washout period)
* Patient suffering from a medical condition prohibiting blood flow occlusion in both arms

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with chest pain and non-obstructive coronary artery disease (20-70% diameter luminal narrowing) will be enrolled in the study 2-30 days following the coronary angiograms
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
MACE | 3 years
  Time to the first occurrence of death, cardiovascular death, non-fatal myocardial infarction, stroke, transient ischemic attack, coronary revascularization, or hospitalization for congestive heart failure.

SECONDARY OUTCOMES:
Rehospitalization for chest pain | 3 years
quality of life questionnaire | 3years
time to the first occurrence of cardiovascular death | 3 years
myocardial infarction | 3 years
Stroke | 3 years
time to the first occurrence of death from any cause | 3 years
hospitalization for worsening heart failure | 3 years
time to the first occurrence of ischemic fatal or non-fatal stroke or transient ischemic attack. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, M.D; Prof, Principal Investigator — Mayo Clinic
Locations (2):
- Israel (2):
  - Meir Hospital, Kfar Saba
  - Tel Hashomer, Ramat Gan

IPD SHARING:
Plan to Share IPD: Undecided